CLINICAL TRIAL: NCT06309043
Title: A Randomized, Single Intravenous Dose, Parallel Phase I Clinical Study to Compare the Pharmacokinetic Characteristics, Safety, and Immunogenicity of HLX05 Vs. Erbitux® (Cetuximab) in Healthy Adult Male Chinese Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX05-001
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: EGFR Overexpression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HLX05 (Experimental)
  Interventions: Drug: recombinant anti-EGFR human/murine chimeric monoclonal antibody injection
- EU-sourced Erbitux (Active Comparator)
  Interventions: Drug: recombinant anti-EGFR human/murine chimeric monoclonal antibody injection
- US-sourced Erbitux (Active Comparator)
  Interventions: Drug: recombinant anti-EGFR human/murine chimeric monoclonal antibody injection
- CN-sourced Erbitux (Active Comparator)
  Interventions: Drug: recombinant anti-EGFR human/murine chimeric monoclonal antibody injection

INTERVENTIONS:
Drug: recombinant anti-EGFR human/murine chimeric monoclonal antibody injection — a single dose，250 mg/m2

SUMMARY:
This is a randomized, single intravenous dose, parallel study to compare the PK characteristics, safety, tolerability, and immunogenicity of HLX05 vs. Erbitux® (US-, EU-, and CN-sourced) in healthy adult male Chinese subjects. This study is divided into two parts.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males aged 18-50 years (inclusive); 2. Body mass index (BMI) = body weight (kg)/height2 (m2); BMI between 18.5 and 28.0 (inclusive), and body weight of male subjects ≥ 50 kg; 3. Subjects without abnormalities or those with abnormalities with no clinical significance in terms of vital signs measurement, physical examination, clinical laboratory tests (hematology, urinalysis, serum chemistry, infectious disease indicators, coagulation function, cardiac markers, alcohol screening, drug screening, etc.), 12-lead ECG examination, chest X-ray, and abdominal B ultrasound; 4. Subjects who voluntarily take effective contraceptive measures and have no sperm donation plan during the screening period and within 3 months after drug administration, and voluntarily take non-drug contraceptive measures during the trial; 5. After fully understanding the content of the trial and possible adverse reactions, the subjects who voluntarily participate in the trial, are willing to sign the informed consent form (ICF), and are able to complete the study in accordance with the trial protocol.

Exclusion Criteria:

1. With allergic constitution, or history of food or drug allergy; known history of allergy to any ingredient of the study drug or excipients or monoclonal antibody agents; history of infusion reactions;
2. Subjects with a history of cardiovascular, respiratory, endocrine, hepatic, renal, gastrointestinal, nervous system, or hematological, immunological, psychiatric, metabolic obvious abnormalities, skin diseases, or other significant diseases, and are judged by the investigator as unsuitable for participating in the trial;
3. Those with hereditary bleeding tendency or coagulation disorder, or a history of thrombosis or bleeding disorders;
4. With known or suspected history of keratitis, ulcerative keratitis, or severe dry eye disease;
5. With a history of surgery within 3 months prior to screening, or planned surgery during the trial;
6. Intolerant to venipuncture or with a history of needle or blood phobia;
7. With a history of drug abuse within 6 months prior to screening;
8. Use of narcotics within 3 months prior to screening;
9. Subjects who have donated blood including blood components or lost blood (≥ 200 mL), received blood transfusion, or used blood products within 3 months prior to screening;
10. Subjects who have received anti-EGFR targeted drugs (including monoclonal antibodies and TKIs) or other monoclonal antibodies within 3 months prior to screening;

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 268 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
AUC0-inf | 0 to Day 29
  Area under the serum concentration-time curve from time 0 to infinity

SECONDARY OUTCOMES:
Cmax | 0 to Day 29
  Maximum serum concentration
Tmax | 0 to Day 29
  Time to reach maximum serum concentration
CL | 0 to Day 29
  Total clearance
λz | 0 to Day 29
  Apparent terminal elimination rate constant

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No